CLINICAL TRIAL: NCT03552341
Title: Assessing Iodine Status and Associated Health Outcomes in British Women During Pregnancy
Brief Title: Iodine Status in Pregnancy and Associated Health Outcomes
Acronym: Hiba
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: Bradford Teaching Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Darren Greenwood, Senior Lecturer in Biostatistics, University of Leeds
Other Study IDs: PR-R10-0514-11004
Record Dates: First submitted 2018-05-11; First posted 2018-06-11 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Cognitive Developmental Delay; Birth Weight
Keywords: Iodine; Cognitive function; Birth outcomes; Pregnancy
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 7000 urine samples from the Born in Bradford cohort. 200 urine and blood samples during pregnancy and lactation from the Hiba longitudinal cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Maternal iodine status — Urinary iodine concentration during pregnancy at 26 weeks' gestation (Bord in Bradford study) and at 12, 26 and 36 weeks' gestation, 6, 18 and 30 weeks postpartum (Hiba longitudinal study). This is primarily in the form of Iodine to Creatinine ratio, to take spot urine volume into account. There is no intervention in this observational study.

SUMMARY:
Iodine is a key micronutrient in the diet, essential for healthy growth, and is particularly important during pregnancy and breastfeeding when demands are increased to support the developing baby. Many people are thought to lack all the iodine they need, and this is a greater issue during and shortly after pregnancy when the body's iodine requirements are greatest. Iodine deficiency complications are potentially serious for both mother and child. Iodine deficiency can lead to thyroid enlargement, lower production of important hormones produced by the thyroid, pregnancy complications in the mother, and impaired growth and developmental problems in babies and children. This research will focus on providing an up-to-date estimate of how many pregnant women do not have enough iodine, and what different levels of iodine might mean in terms of health risks during pregnancy and for childhood development. The investigators will investigate how iodine levels vary over the course of pregnancy and lactation, how this is affected by diet, associated changes in thyroid size and function, and what levels of iodine are linked with greater risk of subsequent health problems. The research will take advantage of existing urine samples collected from mothers during pregnancy in the Born in Bradford birth cohort study, where the investigators also know of any adverse pregnancy outcomes, as well as any developmental problems for the baby and in early childhood.

DETAILED DESCRIPTION:
Background: Pregnant women may be particularly vulnerable to iodine deficiency as requirements increase to support fetal development. There is limited information concerning how maternal iodine status changes during pregnancy. Severe iodine deficiency is associated with deleterious health outcomes during pregnancy including gestational diabetes, preeclampsia, stillbirth, and increased mortality. For the fetus, severe iodine deficiency results in reduced birthweight, increased mortality and neurodevelopmental issues. Several studies suggest 40% of pregnant mothers in the United Kingdom (UK) may not meet the World Health Organization (WHO) definition of iodine sufficiency. Although the effects of severe iodine deficiency are known, the impact of mild-to-moderate deficiencies on maternal health and associated fetal and childhood development are not well understood.

Aims:

1. To provide up-to-date information on iodine status in pregnant women in the UK, including changes during pregnancy and lactation, and the role of diet.
2. To quantify any associations between iodine status during pregnancy, pregnancy outcomes, and cognitive and motor development of the child.
3. To compare the iodine status of mothers in the Born in Bradford cohort to a more nationally representative sample.

Research plan and methods: The investigators will utilize the Born in Bradford (BiB) birth cohort which recruited over 12000 pregnant women between 2007- 2009, and has deposited in a biobank 6971 spot urine samples collected at 26-28 weeks gestation.

Data are available on health outcomes during pregnancy including gestational diabetes, preeclampsia, blood pressure, length of gestation, mortality, mental health. Child outcome measures at birth include weight, length, head circumference, small-for-gestational-age. Childhood developmental measures include height, weight, growth trajectories, motor skills, literacy, numeracy and mental health (Strengths and Difficulties Questionnaire, SDQ). Linkage with educational outcomes has been achieved, including Early Years Foundation Stage (EYFS) outcomes and Standard Assessment Tests (SATS) at both Key Stage 1 (KS1) and Key Stage 2 (KS2).

The investigators will measure all maternal urine samples in BiB to allow sufficient power to detect potential modest-sized associations. This will be conducted using Inductively Coupled Plasma Mass Spectrometry (ICPMS). All maternal baseline characteristics and associated outcome data are available for extraction from the primary BiB database.

The investigators will apply multiple logistic regression and multiple linear regression to ascertain potential associations between maternal iodine status and health and developmental outcomes. Cubic splines will be used to model any nonlinear dose-response associations, making no assumptions regarding any predefined thresholds.

The investigators will also conduct a longitudinal substudy to ascertain how iodine status varies between trimesters (The Hiba study). 200 pregnant women will be recruited at 12 week dating scans and the following collected: baseline characteristics, urine samples for iodide analysis, blood for thyroid stimulating hormone (TSH), free thyroxine (fT4) and triiodothyronine (fT3), thyroglobulin, Glomerular Filtration Rate (GFR) based on serum creatinine, visual inspection of the thyroid using standard methods, dietary intake using a validated online 24h recall tool (myfood24). Data collection will be repeated at 26 and 36 weeks' gestation, and 6, 18 and 30 weeks postpartum. The proposed substudy will clarify how iodine status alters in pregnancy and lactation, and any associated thyroid hormone changes. The investigators will identify key sources of iodine in the diet and ascertain dietary patterns associated with different iodine status. To compare results to a more nationally representative sample, spot urines will be analysed from approximately 650 women in the SCOPE birth-cohort (London, Leeds and Manchester).

ELIGIBILITY:
Inclusion criteria:

* Female (Both Born in Bradford and Hiba longitudinal cohorts)
* Able to provide informed consent (Both Born in Bradford and Hiba longitudinal cohorts)
* Confirmed pregnant at 26-28 week Oral Glucose Tolerance Test (OGTT) (Born in Bradford cohort)
* Confirmed 9-15 weeks pregnant at 12 week dating scan (Hiba longitudinal cohort)
* Aged 18-40 years (Hiba longitudinal cohort)
* No medical or known first degree family history of a thyroid condition (Hiba longitudinal cohort).

Exclusion criteria:

* Inability to provide informed consent (Both Born in Bradford and Hiba longitudinal cohorts)
* Current or former medical history of thyroid disease (Hiba longitudinal cohort)
* Use of thyroid related medications (Hiba longitudinal cohort)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The Born in Bradford cohort profile is published here: [doi:10.1093/ije/dys112] All women booked for delivery at the Bradford Royal Infirmary at 26-28 weeks gestation. All of the recruited women who provided urine samples are included in our Born in Bradford analysis.
  The Hiba longitudinal study replicates this process, but at the 12 week dating scan.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Born in Bradford: Early Years Foundation Stage (EYFS) profiles | Ages 3 to 5
  The EYFS average points total over 17 domains (score range 17 to 41) and summarised using achievement of Good Level of Development (GLD) (binary).

SECONDARY OUTCOMES:
Born in Bradford: Key Stage 1 (KS1) educational outcomes | Ages 5 to 8
  Year 1 phonics screening test (score range 0 to 40) and KS1 SATS scores in Reading, Writing, Mathematics and Science (working securely at level 2b or beyond pre-2016 or working at the expected standard or beyond for 2016 onwards, binary) will be presented.
Born in Bradford: Letter identification | Ages 3 to 5
  Letter identification (standardised)
Born in Bradford: Receptive vocabulary | Ages 3 to 5
  Receptive vocabulary using the British Picture Vocabulary Scale (BPVS)(standardised)
Born in Bradford: Social functioning | Ages 3 to 5
  Social functioning using the Strengths and Difficulties Questionnaire (SDQ) total difficulty score and split by domains (e.g. internalising and externalising)
Born in Bradford: Fine motor skills | Ages 3 to 5
  Fine motor skills using the Clinical Kinematic Assessment Tool (CKAT) overall battery score, along with Tracking, Aiming and Tracing CKAT sub-scores.
Born in Bradford: Birth weight centile | At birth
  The main birth outcome of interest is birth weight centile, calculated using the version 8.0.1 of the Bulk centile calculator provided by the Gestation Network based at the Perinatal Institute for Maternal and Child Health
Born in Bradford: Apgar score | At 1 minute and 5 minutes after birth.
  Apgar score (ordinal).
Born in Bradford: Diagnosis of autism | Up to age 11.
  Confirmed diagnosis of autism based on Read codes in linked General Practitioner records.
Born in Bradford: Diagnosis of attention deficit hyperactivity disorder (ADHD) | Up to age 11.
  Confirmed diagnosis of attention deficit hyperactivity disorder (ADHD) based on Read codes in linked General Practitioner records.
Hiba longitudinal study: Urinary iodine status | 12, 26 and 36 weeks' gestation during pregnancy, and 6, 18 and 30 weeks' postpartum.
  The main outcome of interest is urinary iodine status (primarily in the form of iodine to creatinine ratio to take account of spot urine volumes) changes during pregnancy and lactation (continuous)
Hiba longitudinal cohort: thyroid stimulating hormone (TSH) | 12, 26 and 36 weeks' gestation during pregnancy, and 6, 18 and 30 weeks' postpartum.
  Changes in thyroid stimulating hormone (TSH) during gestation and lactation.
Hiba longitudinal cohort: triiodothyronine (fT3) | 12, 26 and 36 weeks' gestation during pregnancy, and 6, 18 and 30 weeks' postpartum.
  Changes in triiodothyronine (fT3) during gestation and lactation.
Hiba longitudinal cohort: free thyroxine (fT4) | 12, 26 and 36 weeks' gestation during pregnancy, and 6, 18 and 30 weeks' postpartum.
  Changes in free thyroxine (fT4) during gestation and lactation.
Hiba longitudinal cohort: thyroglobulin | 12, 26 and 36 weeks' gestation during pregnancy, and 6, 18 and 30 weeks' postpartum.
  Changes in thyroglobulin during gestation and lactation.
Hiba longitudinal cohort: thyroid size | 12, 26 and 36 weeks' gestation during pregnancy, and 6, 18 and 30 weeks' postpartum.
  Changes in thyroid size, measured by palpation, using a standard protocol, during gestation and lactation.
Hiba longitudinal cohort: maternal dietary iodine intake (micrograms) | 12, 26 and 36 weeks' gestation during pregnancy, and 6, 18 and 30 weeks' postpartum.
  Identification of highest ranking food items in terms of contribution to iodine in the maternal diet as measured using the myfood24 tool

OTHER OUTCOMES:
Born in Bradford: length of gestation | At birth
  length of gestation (weeks), presenting pre-term delivery (<37 weeks)
Born in Bradford: congenital anomalies | At birth
  Diagnosis of congenital anomalies from linked congenital anomalies records (binary)
Born in Bradford: childhood growth trajectories | From 26 weeks gestation, through to age 11
  Childhood growth trajectories (weight in kg)
Born in Bradford: Key Stage 2 (KS2) educational outcomes | Ages 8 to 11
  Key Stage 2 (KS2) SATS scores in English grammar, punctuation and spelling, English reading, and Mathematics.
Born in Bradford: maternal mental health | From 26 weeks gestation, through to age 11
  Patient Health Questionnaire 9 (PHQ-9) depression test questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Darren C Greenwood, PhD, Principal Investigator — University of Leeds; Laura J Hardie, PhD, Principal Investigator — University of Leeds

IPD SHARING:
Plan to Share IPD: Yes
Born in Bradford welcomes collaboration with other researchers. The BiB website has details of how to submit expressions of interest and has short proformas for these. All suggestions will be reviewed by the BiB Executive Group on a monthly basis, and we aim to get back to potential collaborators within 8 weeks.
Time Frame: Ongoing.
Access Criteria: Submit expressions of interest on a short proforma. All suggestions will be reviewed by the BiB Executive Group.
URL: https://borninbradford.nhs.uk/

REFERENCES:
- [Result] Snart CJP, Keeble C, Taylor E, Cade JE, Stewart PM, Zimmermann M, Reid S, Threapleton DE, Poston L, Myers JE, Simpson NAB, Greenwood DC, Hardie LJ. Maternal Iodine Status and Associations with Birth Outcomes in Three Major Cities in the United Kingdom. Nutrients. 2019 Feb 20;11(2):441. doi: 10.3390/nu11020441. PMID 30791590
- [Result] Snart CJP, Threapleton DE, Keeble C, Taylor E, Waiblinger D, Reid S, Alwan NA, Mason D, Azad R, Cade JE, Simpson NAB, Meadows S, McKillion A, Santorelli G, Waterman AH, Zimmermann M, Stewart PM, Wright J, Mon-Williams M, Greenwood DC, Hardie LJ. Maternal iodine status, intrauterine growth, birth outcomes and congenital anomalies in a UK birth cohort. BMC Med. 2020 Jun 11;18(1):132. doi: 10.1186/s12916-020-01602-0. PMID 32522280
- [Result] Threapleton DE, Snart CJP, Keeble C, Waterman AH, Taylor E, Mason D, Reid S, Azad R, Hill LJB, Meadows S, McKillion A, Alwan NA, Cade JE, Simpson NAB, Stewart PM, Zimmermann M, Wright J, Waiblinger D, Mon-Williams M, Hardie LJ, Greenwood DC. Maternal iodine status in a multi-ethnic UK birth cohort: Associations with child cognitive and educational development. Paediatr Perinat Epidemiol. 2021 Mar;35(2):236-246. doi: 10.1111/ppe.12719. Epub 2020 Sep 1. PMID 32870514
- [Result] Threapleton DE, Waiblinger D, Snart CJP, Taylor E, Keeble C, Ashraf S, Bi S, Ajjan R, Azad R, Hancock N, Mason D, Reid S, Cromie KJ, Alwan NA, Zimmermann M, Stewart PM, Simpson NAB, Wright J, Cade JE, Hardie LJ, Greenwood DC. Prenatal and Postpartum Maternal Iodide Intake from Diet and Supplements, Urinary Iodine and Thyroid Hormone Concentrations in a Region of the United Kingdom with Mild-to-Moderate Iodine Deficiency. Nutrients. 2021 Jan 14;13(1):230. doi: 10.3390/nu13010230. PMID 33466826
- [Result] Cromie KJ, Threapleton DE, Snart CJP, Taylor E, Mason D, Wright B, Kelly B, Reid S, Azad R, Keeble C, Waterman AH, Meadows S, McKillion A, Alwan NA, Cade JE, Simpson NAB, Stewart PM, Zimmermann M, Wright J, Waiblinger D, Mon-Williams M, Hardie LJ, Greenwood DC. Maternal iodine status in a multi-ethnic UK birth cohort: associations with autism spectrum disorder. BMC Pediatr. 2020 Dec 5;20(1):544. doi: 10.1186/s12887-020-02440-y. PMID 33276760
- Available data/document: Individual Participant Data Set — https://borninbradford.nhs.uk/ — Submit expressions of interest on a short proforma. All suggestions will be reviewed by the BiB Executive Group.

DOCUMENTS (3):
  • Statistical Analysis Plan (2018-11-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT03552341/SAP_003.pdf
  • Informed Consent Form: Born in Bradford cohort Informed Consent Form (2010-07-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT03552341/ICF_001.pdf
  • Informed Consent Form: Hiba longitudinal cohort Informed Consent Form (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03552341/ICF_002.pdf